CLINICAL TRIAL: NCT01059708
Title: Outcome Following Carbon Monoxide Poisoning in Children
Acronym: CO PED
Status: Terminated | Type: Observational
Why Stopped: Low enrollment.
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Deseret Foundation (Other)
Responsible Party: Susan K. Churchill, APRN-NP, Clinical Coordinator, Intermountain Healthcare
Other Study IDs: 1004920
Record Dates: First submitted 2010-01-28; First posted 2010-02-01 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Carbon Monoxide Poisoning
Keywords: outcomes carbon monoxide poisoning children pediatric
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be obtained by mouthwash, spit collection, or buccal swab,
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CO poisoned children: Children, ages 6-16, who have been poisoned by carbon monoxide

SUMMARY:
Carbon monoxide poisoning is common. Many adults with CO poisoning have long-term, even permanent brain injury following poisoning. However, very little is known about the long-term outcome of children with carbon monoxide (CO) poisoning. In this study we plan to perform cognitive (thinking) and vestibular (balance) testing in children (ages 6 to 16)at 6 weeks and 6 months following CO poisoning.

At the 6-week visit, if the child and parents agree, we will ask each child to provide a DNA sample by one of three methods: mouthwash, spit collection, or swabbing the inside of the child's cheek. Each child's DNA will be analyzed for genes that are known to affect outcome following brain injury.

DETAILED DESCRIPTION:
Each child's participation in this study is expected to last 6 months. Testing will be scheduled around 6 weeks after the carbon monoxide (CO) poisoning episode. During testing, each child will be asked to complete tests that measure cognitive (thinking), emotional, and behavioral performance. We will collect information from each child's medical record about the CO poisoning episode, and we will have a parent complete a questionnaire about any problems he or she may have observed in their child since the poisoning. The cognitive testing will take about 3.5 hours at the 6-week interval, and 2.5 hours at the 6-month interval.

Around the same time, each child will also be scheduled for vestibular (balance) testing at the Intermountain Hearing and Balance Center. Vestibular testing will occur twice, at 6-weeks and 6-months following poisoning.

At the 6-week visit, if the child and parents agree, we will ask each child to provide a DNA sample by one of three methods: mouthwash, spit collection, or swabbing the inside of the child's cheek. Each child's DNA will be analyzed for genes that are known to affect outcome following brain injury such as apolipoprotein E, and the sample will also be stored for an indefinite period of time. If discoveries are made about other genes that affect outcome following brain injury, each child's DNA will be analyzed for those genes as well.

The primary outcome measure will be the percentage of patients with cognitive sequelae (thinking complications or results) at 6 weeks and 6 months following CO poisoning.

Secondarily, we will also determine:

1. Which individual neurocognitive (thinking) outcomes at 6 weeks and 6 months differ from normative data.
2. Whether there is a difference in neurocognitive (thinking) outcomes between measurement at 6 weeks and 6 months.
3. If there is a difference in the vestibular (balance) health of patients between measurements at 6 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 through 16.
2. Acute carbon monoxide poisoning. Since we will be identifying potentially eligible patients using an electronic tool, the diagnosis of CO poisoning should be established by the evaluating physician. However, with the initial contact with the patients' parents, we will confirm the diagnosis, and only those patients with CO poisoning will be eligible.
3. Willing to come to Salt Lake City or Provo for evaluation

Exclusion Criteria:

1. Prior history of neurological injury with permanent sequelae.
2. Prior history of chronic neurological disorder such as attention deficit disorder, learning disability, multiple sclerosis, cerebral palsy, demyelinating disease, meningitis with sequelae
3. Insulin dependent diabetes (due to the confound of possible brain microvascular disease and episodes of hypoglycemia)
4. Use of illicit drugs
5. Use of alcohol in excess
6. Pregnancy
7. Carbon monoxide poisoning from a suicide attempt or concomitant smoke inhalation
8. Subject or parent/guardian non-English-speaking

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, ages 6-16, following CO poisoning
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with cognitive sequelae at 6 weeks and 6 months following CO poisoning will be reported. | 6 weeks and 6 months after carbon monoxide poisoning incident.

SECONDARY OUTCOMES:
To determine which individual neurocognitive outcomes at 6 weeks and 6 months differ from normative data. | 6 weeks and 6 months after carbon monoxide poisoning incident.
To determine whether there is a difference in neurocognitive outcomes between measurement at 6 weeks and 6 months. | 6 weeks and 6 months after carbon monoxide poisoning incident.
To determine if there is a difference in the vestibular health of patients between measurements at 6 weeks and 6 months. | 6 weeks and 6 months after carbon monoxide poisoning incident.

CONTACTS AND LOCATIONS:
Overall Officials: Lindell K Weaver, MD, Study Director — Intermountain Healthcare, LDSH Hyperbaric Medicine; Susan Churchill, APRN-NP, Principal Investigator — Intermountain Healthcare, LDSH Hyperbaric Medicine
Locations (1):
- Intermountain Healthcare, LDS Hospital, Salt Lake City, Utah, United States